CLINICAL TRIAL: NCT01183741
Title: Clinical Evaluation of the Sotera VisiTM System for Measurement of Systolic and Diastolic Blood Pressures in Adults
Brief Title: Accuracy of Non-Invasive Blood Pressure Measurement in Adults
Acronym: NIBP
Status: Withdrawn | Type: Observational
Sponsor: Sotera Wireless, Inc. (Industry)
Responsible Party: Gary Manning, Vice President Clinical Affairs and Business Development, Sotera Wireless, Inc.
Other Study IDs: SOW-US10-003; 0-00026
Record Dates: First submitted 2010-08-13; First posted 2010-08-18 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension; Hypotension
Keywords: Hypertension; Hypotension; Blood pressure
MeSH Terms: conditions — Hypertension; Hypotension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the accuracy of the Sotera ViSi, an investigational device, to auscultation (measurement with a cuff) in determining systolic and diastolic blood pressure (BP) in adult subjects.

DETAILED DESCRIPTION:
This study is a single-center blinded study that will enroll approximately 150 adult subjects. Trained auscultators will perform the standard auscultation BP measurements. They will be blinded to each other's measurements and from the ViSi measurements.

The study population will be randomized into two groups based on the side of the blood pressure measurement: the left arm group (LAG) and the right arm group (RAG).

The randomization ratio of the LAG and RAG will be 1:1. There will be forced stratification in order to ensure that the study subjects meet the required arm circumference and blood pressure distributions as specified in the SP10:2008 and ISO 81060-2:2009(E) standards.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than 12 years of age at the time of screening.
* Subject's upper arm circumference is between 20cm and 55cm.
* Subject is willing to undergo the Informed Consent process prior to enrollment in the study.
* Subject is willing and able to participate for up to 60 minutes.

Exclusion Criteria:

* Subject is participating in another clinical study that may interfere with the results of this study.
* Subject is unable to have a blood pressure measurement taken from either arm for any reason.
* Subject is evaluated by the Investigator and found to be medically unsuitable for participation in this study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Eligible subjects are adults of any ethnic background who consent to spot-check blood pressure measurements and in whom paired blood pressure measurements with the ViSi will be feasible during a single visit. Subjects need to be greater than 12 years of age on the date of measurement and need to meet all the other inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Drehobl, M.D., Principal Investigator — Scripps Health
Locations (1):
- Scripps Clinic Rancho Bernardo, San Diego, California, United States